CLINICAL TRIAL: NCT01789307
Title: Lactose: A Unique Carbohydrate Enabling Homeostatic Regulation of Blood Glucose & Insulin
Brief Title: Lactose, Sucrose & Corn Syrup Tolerance
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of British Columbia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double
Other Study IDs: H12-01647
Record Dates: First submitted 2012-12-20; First posted 2013-02-12 (Estimated); Last update posted 2014-07-04 (Estimated); Status verified 2014-07

CONDITIONS: Focus of Study: Oral Tolerance Test With Glucose, Lactose, Sucrose
MeSH Terms: interventions — High Fructose Corn Syrup; Sucrose

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- corn syrup solids (Active Comparator): corn syrup solids oral ingestion
  Interventions: Dietary Supplement: corn syrup solids
- sucrose (Experimental): sucrose oral ingestion
  Interventions: Dietary Supplement: sucrose

INTERVENTIONS:
Dietary Supplement: corn syrup solids — oral ingestion 50 grams, 2 doses
  Other Names: corn syrup
  Arms: corn syrup solids
Dietary Supplement: sucrose — oral ingestion 50 grams, 2 doses
  Arms: sucrose

SUMMARY:
Lactose, one of the key nutrients in human milk may be critically important to infants for more reasons than being a source of energy. We are interested in understanding how lactose when compared to other sugars influences how nutrients, specifically macronutrients are handled after digestion and absorption. To date, there have been no studies looking at how fat and protein varies when lactose compared to other sugars is ingested. There may be metabolic advantages to considering lactose for nutrition support of premature infants rather than glucose or dextrose as is often used in intravenous feeds, or the corn syrup solids in lactose-free formulas. We hope the information from this study will provide new information on the unique aspects of lactose.

Hypothesis: The hypothesis is that providing carbohydrate as lactose:

1. minimizes the amount of carbohydrate that is converted into fat
2. enables a relatively constant metabolic state throughout feeding interval that avoids swings of high to low insulin, glucose, and fats.

ELIGIBILITY:
Inclusion Criteria:

* male
* at least 19 years of age
* body mass index (BMI) between 18.5 and 25
* fasting blood glucose level < 6.1 mmol/L (110 mg/dL) measured by glucometer on the day of the study and
* comfortable speaking, reading and understanding English
* comfortable drinking at least one cup (250 ml) of milk
* non-smoking

Exclusion Criteria:

* not willing to provide blood samples, have
* impaired lactose or glucose tolerance,
* pre-diabetes, diabetes mellitus and any other endocrine disorder,
* coronary heart disease, liver function test abnormalities or any chronic disease
* routinely take medications, including aspirin, cyclooxygenase-2 inhibitors, statins and fish oil
* consuming more than 1 alcoholic drink per day

Ages: 19 Years to 60 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2013-01; Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
Postprandial changes in plasma insulin, glucagon, triglycerides and amino acids. | 6 hours
  Area under the curve changes in the outcome measures following oral ingestion.

SECONDARY OUTCOMES:
Postprandial changes in plasma fatty acids. | 6 hours
  Area under the curve analyses of changes in plasma fatty acids following oral ingestion

CONTACTS AND LOCATIONS:
Overall Officials: Sheila M Innis, PhD, Principal Investigator — University of British Columbia, Child & Family Research Institute
Locations (1):
- Child & Family Research Institute, Vancouver, British Columbia, Canada